CLINICAL TRIAL: NCT00715247
Title: Polycythemia Vera, Myelofibrosis and Essential Thrombocythemia: Identification of PV, MF & ET Genes
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Collaborators: Myeloproliferative Disorders-Research Consortium (Network); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 17793; 1P01CA10867101A2 (Other Grant/Funding Number: NCI)
Record Dates: First submitted 2008-07-11; First posted 2008-07-15 (Estimated); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Polycythemia Vera; Essential Thrombocythemia; Myelofibrosis
Keywords: Myeloproliferative Disorders; Hematological Malignancies; Polycythemia Vera; Essential Thrombocythemia; Myelofibrosis; Genetics; Chronic Leukemia
MeSH Terms: conditions — Polycythemia Vera; Thrombocythemia, Essential; Primary Myelofibrosis; Myeloproliferative Disorders; Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood and bone marrow aspirate
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Affected Population: Patients suspected to have one of the following blood disorders: polycythemia vera, myelofibrosis or essential thrombocythemia.
- Healthy Female Controls: Healthy females who do not have the blood disorders; Polycythemia Vera, Essential Thrombocythemia and/or Myelofibrosis.

SUMMARY:
The purpose of this project is to find genes whose mutations cause Polycythemia Vera, Essential Thrombocythemia and Primary Myelofibrosis.

DETAILED DESCRIPTION:
Polycythemia Vera (PV), Essential Thrombocythemia (ET) and Primary Myelofibrosis (PMF), also known as the Philadelphia Chromosome negative myeloproliferative disorders (MPDs), are not congenital, but acquired. The purpose of this project is to find genes whose mutations cause these disorders, as well as improve diagnostic measures for these diseases. When this is accomplished new therapies to control and eventually cure the disease can be designed.

All subjects will be asked to donate 4-6 teaspoons of blood. On occasion, if the blood cells from a particular sample do not grow well and the DNA from that sample is used up or other tests are needed, we may ask to collect additional samples. In patients who have undergone a bone marrow biopsy as part of their clinical evaluation, we will test the reproducibility between pathologists for the revised 2008 WHO diagnostic criteria to diagnose myeloproliferative disorders (MPD).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with an elevated hemoglobin concentration (>18 in males and >16 in females) and who are suspected to have congenital or acquired primary polycythemia
2. Patients with a persistent thrombocytosis (>400,000) that does not have an obvious secondary cause
3. Patients with a bone marrow biopsy that shows increased cellularity and fibrosis
4. Patients where there is clinical concern for primary myelofibrosis, such as anemia in combination with leukocytosis, thrombocytosis, splenomegaly and/or a leukoerythroblastic blood smear
5. Patients with thrombosis at unusual sites, such as Budd-Chiari syndrome, can have early PV before hemoglobin is elevated, these patients will also be included.

Exclusion Criteria:

1. Subjects who have a known acquired cause of polycythemia (increased hemoglobin/hematocrit) such as people living in high altitudes (in excess of 14,000 feet), subjects with heart disease, left to right heart shunt, severe hypoxia or severe pulmonary disease will be excluded from this study.
2. Subjects with a known acquired cause of thrombocytosis.
3. Subjects will be excluded if they cannot demonstrate decision making capacity sufficient to agree or decline the blood drawing or use of their blood for the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients suspected to have one of the following blood disorders: polycythemia vera, myelofibrosis or essential thrombocythemia.
Sampling Method: Non-Probability Sample
Enrollment: 726 (Actual)
Dates: Start 2006-07; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Identify genes whose mutations cause Polycythemia Vera, Essential Thrombocythemia and Primary Myelofibrosis. | Weekly

SECONDARY OUTCOMES:
To determine if there are proteins expressed by cells from patients that might be targets for the immune response. | Weekly

CONTACTS AND LOCATIONS:
Overall Officials: Josef T Prchal, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

REFERENCES:
- [Background] Jelinek J, Li J, Mnjoyan Z, Issa JP, Prchal JT, Afshar-Kharghan V. Epigenetic control of PRV-1 expression on neutrophils. Exp Hematol. 2007 Nov;35(11):1677-83. doi: 10.1016/j.exphem.2007.09.008. PMID 17976520
- [Background] Agarwal N, Mojica-Henshaw MP, Simmons ED, Hussey D, Ou CN, Prchal JT. Familial polycythemia caused by a novel mutation in the beta globin gene: essential role of P50 in evaluation of familial polycythemia. Int J Med Sci. 2007 Oct 4;4(4):232-6. doi: 10.7150/ijms.4.232. PMID 17952198
- [Background] Gaikwad A, Verstovsek S, Yoon D, Chang KT, Manshouri T, Nussenzveig R, Cortes J, Vainchenker W, Prchal JT. Imatinib effect on growth and signal transduction in polycythemia vera. Exp Hematol. 2007 Jun;35(6):931-8. doi: 10.1016/j.exphem.2007.03.012. PMID 17533047
- [Background] Chen GL, Prchal JT. X-linked clonality testing: interpretation and limitations. Blood. 2007 Sep 1;110(5):1411-9. doi: 10.1182/blood-2006-09-018655. Epub 2007 Apr 13. PMID 17435115
- [Background] Gaikwad A, Nussenzveig R, Liu E, Gottshalk S, Chang K, Prchal JT. In vitro expansion of erythroid progenitors from polycythemia vera patients leads to decrease in JAK2 V617F allele. Exp Hematol. 2007 Apr;35(4):587-95. doi: 10.1016/j.exphem.2006.12.007. PMID 17379069
- [Background] Hoffman R, Prchal JT, Samuelson S, Ciurea SO, Rondelli D. Philadelphia chromosome-negative myeloproliferative disorders: biology and treatment. Biol Blood Marrow Transplant. 2007 Jan;13(1 Suppl 1):64-72. doi: 10.1016/j.bbmt.2006.11.003. PMID 17222772
- [Background] Nussenzveig RH, Swierczek SI, Jelinek J, Gaikwad A, Liu E, Verstovsek S, Prchal JF, Prchal JT. Polycythemia vera is not initiated by JAK2V617F mutation. Exp Hematol. 2007 Jan;35(1):32-8. doi: 10.1016/j.exphem.2006.11.012. PMID 17198871
- [Background] Chen GL, Liu E, Naidoo K, Popat U, Coetzer TL, Prchal JT. Idiopathic myelofibrosis without dacryocytes. Haematologica. 2006 Jun;91(6 Suppl):ECR29. PMID 16785132
- [Background] Finazzi G, Gregg XT, Barbui T, Prchal JT. Idiopathic erythrocytosis and other non-clonal polycythemias. Best Pract Res Clin Haematol. 2006;19(3):471-82. doi: 10.1016/j.beha.2005.07.006. PMID 16781484
- [Background] Chen G, Prchal JT. Polycythemia vera and its molecular basis: an update. Best Pract Res Clin Haematol. 2006;19(3):387-97. doi: 10.1016/j.beha.2005.07.003. PMID 16781479
- [Background] Popat U, Frost A, Liu E, Guan Y, Durette A, Reddy V, Prchal JT. High levels of circulating CD34 cells, dacrocytes, clonal hematopoiesis, and JAK2 mutation differentiate myelofibrosis with myeloid metaplasia from secondary myelofibrosis associated with pulmonary hypertension. Blood. 2006 May 1;107(9):3486-8. doi: 10.1182/blood-2005-08-3319. Epub 2006 Jan 17. PMID 16418333
- [Background] Skoda R, Prchal JT. Chronic myeloproliferative disorders--introduction. Semin Hematol. 2005 Oct;42(4):181-3. doi: 10.1053/j.seminhematol.2005.08.004. No abstract available. PMID 16210031